### NCT02320149

## Study SC1401

Title: A Randomized, Multicenter, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of 1.5 mg/kg per Day of Sarecycline Compared to Placebo in the Treatment of Acne Vulgaris.

Protocol Date: December 16, 2015

Statistical Analysis Plan (SAP) Date: March 3, 2017



#### Study SC1401

A Randomized, Multicenter, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of 1.5 mg/kg per Day of Sarecycline Compared to Placebo in the Treatment of Acne Vulgaris

#### STATISTICAL ANALYSIS PLAN – Amendment 1

Final: 20 Feb 2017

Revised: 03 Mar 2017 (Amendment 1 Date)

#### **Confidentiality Statement**

The following contains confidential, proprietary information which is the property of Allergan, Inc. and may not, in full or part, be passed on, reproduced, published, distributed to any person, or submitted to any regulatory authority without the express written permission of Allergan, Inc.

| <u>2.0</u> | | <u> 1</u> A | ABLE OF CONTENTS | |
|---|---|---|---|---|
| 1.0 | TITLE | PAGE | | 1 |
| 2.0 | TABL | E OF CO | NTENTS | 2 |
| 3.0 | LIST | OF ABBR | EVIATIONS | 4 |
| 4.0 | INTRO | DUCTIO | N | 5 |
| 5.0 | OBJEC | CTIVES | | 9 |
| 6.0 | ANAL<br>6.1<br>6.2<br>6.3<br>6.4 | SCREE<br>SAFET<br>INTEN | PULATIONS AND DATASETS<br>NED POPULATIONY POPULATION<br>T-TO-TREAT POPULATION<br>ROTOCOL POPULATION | 10<br>10 |
| 7.0 | SUBJE | ECT DISP | OSITION | 12 |
| 8.0 | DEMO | GRAPHI | CS AND OTHER BASELINE CHARACTERISTICS | 13 |
| 9.0 | 9.1<br>9.2 | EXTEN | RPOSURE AND TREATMENT COMPLIANCET OF EXPOSURE | 15 |
| 10.0 | 10.1<br>10.2<br>10.3<br>10.4<br>10.5 | CO-PR<br>10.1.1<br>10.1.2<br>SECON<br>ADDIT<br>SUBGE<br>OTHER<br>10.5.1<br>10.5.2<br>ADDIT | IONAL EFFICACY ANALYSES | |
| 11.0 | SAFET<br>11.1<br>11.2<br>11.3<br>11.4<br>11.5 | ADVER<br>CLINIC<br>VITAL<br>ELECT<br>OTHER | YSES | 23 24 25 26 27 |
| 12.0 | HEAL | TH OUT | COMES ANALYSES | 28 |
| 13.0 | INTER | ANA MIS | LYSIS | 29 |
| 14.0 | DETE | RMINAT | ION OF SAMPLE SIZE | 30 |

| 15.0 | STATI | STICAL | SOFTWARE | 31 |
|---|---|---|---|---|
| 16.0 | DATA | | ING CONVENTIONS | |
| | 16.1 | VISIT 7 | ΓΙΜΕ WINDOWS | 32 |
| | 16.2 | MISSIN | NG DATA HANDLING FOR PRIMARY AND SECONDARY EFFICACY | |
| | | ENDPO | DINTS | 32 |
| | 16.3 | REPEA | TED OR UNSCHEDULED ASSESSMENTS OF SAFETY PARAMETERS | 334 |
| | 16.4 | MISSIN | NG DATE OF THE LAST DOSE OF INVESTIGATIONAL PRODUCT | 35 |
| | 16.5 | MISSIN | NG SEVERITY ASSESSMENT FOR ADVERSE EVENTS | 35 |
| | 16.6 | MISSIN | NG RELATIONSHIP TO INVESTIGATIONAL PRODUCT FOR | |
| | | ADVE | RSE EVENTS | 35 |
| | 16.7 | MISSIN | NG DATE INFORMATION FOR ADVERSE EVENTS | 35 |
| | 16.8 | Missing | Date Information for Prior or Concomitant Medications | 36 |
| | | 16.8.1 | Incomplete Start Date | 36 |
| | | | Incomplete Stop Date | |
| | 16.9 | | ACTER VALUES OF CLINICAL LABORATORY PARAMETERS | |
| 17.0 | CHAN | GES IN A | AMENDMENT 1 OF THE STATISTICAL ANALYSIS PLAN | 40 |
| 18.0 | REFE | RENCES | | 41 |
| 19.0 | | | Conventional US Reporting of Reference Ranges for Clinical Laboratory | 42 |
| | | Evaluat | ions | 42 |

#### 3.0 LIST OF ABBREVIATIONS

AE adverse event

ANCOVA analysis of covariance
CFB change from baseline
CI confidence interval

CMH Cochran-Mantel-Haenszel

CRF case report form

ECG electrocardiogram, electrocardiographic

IGA Investigator's Global Assessment
IRT Interactive Response Technology

ITT intent to treat

LOCF last observation carried forward

MI multiple imputation

MMRM mixed model repeated measures

OC observed cases

PCS potentially clinically significant

QTc QT interval corrected for heart rate

QTcB QT interval corrected for heart rate using the Bazett formula

 $(QTcB = QT/(RR)^{\frac{1}{2}})$ 

QTcF QT interval corrected for heart rate using the Fridericia formula

 $(QTcF = QT/(RR)^{1/3})$ 

SAE serious adverse event SAP statistical analysis plan

SI Le Système International d'Unités (International System of Units)

SID subject identification number

TEAE treatment-emergent adverse event

#### 4.0 INTRODUCTION

This statistical analysis plan (SAP) provides a more technical and detailed elaboration of the statistical analyses of the efficacy and safety data as outlined and/or specified in the final protocol of Study SC1401 (15 Aug 2014) and the most recent amendment (Version 3 dated 16 Dec 2015).

Specifications of tables, figures, and data listings are contained in a separate document. The SAP for pharmacokinetic/pharmacodynamic data will be prepared separately.

Study SC1401 is a phase 3 multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate efficacy and safety of an approximate 1.5 mg/kg/day dose of oral sarecycline compared to placebo in the treatment of moderate to severe facial acne vulgaris. The study will include approximately 1000 males and females 9 to 45 years of age with moderate to severe facial acne vulgaris and no disorders that would preclude the use of tetracycline-class antibiotics at approximately 50 sites.

The study includes a screening period of up to 35 days to establish eligibility and baseline conditions followed by a 12-week treatment period. Eligible subjects will be randomized in a 1:1 ratio to receive daily oral doses of either 1.5 mg/kg sarecycline tablets or placebo tablets. Subjects will return to the clinic on an outpatient basis following 3, 6, 9 and 12 weeks of treatment. At each clinic visit, facial acne will be evaluated through lesion counts and Investigator's Global Assessment (IGA) scores by visual inspection; non-facial inflammatory acne will also be evaluated by IGA of the neck, chest and back. The co-primary efficacy endpoints of the study are the absolute change from baseline in the facial inflammatory lesion count at Week 12 and a dichotomized IGA (dichotomized to reflect either 'success' or 'failure' with 'success' defined as at least a 2-point decrease from baseline in the IGA assessment and a score of clear [0] or almost clear [1] on the IGA assessment) at Week 12. Safety evaluations (adverse events, vital signs, clinical laboratory evaluations, electrocardiograms (ECG) and physical examinations) will be conducted at specific treatment period visits and at study termination.

The study drug, referred to as investigational product in this statistical analysis plan, quantity and dispensing schedule for this study are as follows:

| Visit | Quantity Dispensed |
|---------------------|--------------------|
| Screen Visit (SV) 2 | 30 |
| 1 | 30 |
| 2 | 30 |
| 3 | 30 |

The schedule of evaluations for Study SC1401 is presented in Table 4-1.

Table 4-1. Study Schedule of Events: Study SC1401

| Table 4-1. | Screening Period Treatment Period | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | ening Period | Televitor | ¥72.24 4 | | | X72-24 4 | <b>X</b> 72 |
| | SV1 | SV2 | Telephone<br>Contact | Visit 1<br>Week 3 | Visit 2<br>Week 6 | Visit 3<br>Week 9 | Visit 4<br>Week 12 | Visit 5 <sup>d</sup> |
| | | (Baseline | Week 1 | | | | | Week 13 |
| | | Assessment) | ± 3 d | ± 3 d | ± 3 d | ± 3 d | /ET<br>± 3 d | /ET<br>± 3 d |
| T.C. 1 | | | ±3 u | | | | ± 3 u | ±30 |
| Informed | X | | | | | | | |
| Consent | | | | | | | | |
| Assign Subject<br>Number using | X | | | | | | | |
| the IRT | | | | | | | | |
| Inclusion/<br>Exclusion | X | X | | | | | | |
| Demographic<br>Data | X | | | | | | | |
| Medical/<br>Surgical<br>History | X | | | | | | | |
| Physical<br>Examination | X | Xª | | | | | X | X |
| Height &<br>Weight | X | Weight<br>only | | | | | Weight only | Weight only |
| Vital Signs | X | X | | X | X | X | X | X |
| Hematology,<br>Serum<br>Chemistry,<br>Urinalysis and<br>Lipids | X | X <sup>b</sup> | | X | | | Х | |
| TSH, Free T4<br>and T3 | X | | | | | | X | |
| Urine pregnancy test | X | X | | X | X | X | X | X |
| ECG | X | | | | | | X | |
| Facial<br>Investigator's<br>Global<br>Assessment | | X | | X | X | X | X | |
| Facial Lesion<br>Counts | | X | | X | X | X | X | |
| Facial<br>Photographs | | X | | X | X | X | X | |
| Non-facial<br>Investigator's<br>Global<br>Assessment | | X | | X | X | X | X | |

Table 4–1. Study Schedule of Events: Study SC1401

| 1 4016 4-1. | | ening Period | ning Period Treatment Period | | | | | |
|---|---|---|---|---|---|---|---|---|
| | SV1 | SV2 | | | | | | Visit 5 <sup>d</sup> |
| | 311 | (Baseline | Contact | Week 3 | Week 6 | Week 9 | Week 12 | Week 13 |
| | | Assessment) | Week 1 | ±3 d | ±3d | ±3d | /ET | /ET |
| | | rissessment | ± 3 d | ±5 <b>u</b> | ± 5 <b>u</b> | ± 5 u | ± 3 d | ± 3 d |
| Skindex<br>Questionnaire | | X | | | | | X | |
| Dispense Diary<br>for Subjects<br>Participating in<br>PK Sampling | | X | | | | X | | |
| PK Blood<br>Sample<br>Collection for<br>PK 1, PK 2,<br>and PK 3 <sup>c</sup> | | | | X | | | X | |
| Review and<br>Collect Diaries | | | | X | | | X | |
| Randomization | | X | | | | | | |
| Dispense<br>Study drug | | X | | X | X | X | $\mathbf{X}^{\mathbf{d}}$ | |
| Study drug<br>Accountability<br>/Compliance | | | X | X | X | X | X | |
| Concomitant<br>Medication<br>Use | X | X | | X | X | X | X | X |
| Adverse<br>Events | X | X | X | X | X | X | X | X |

ECG= electrocardiogram; ET= End of treatment; X<sup>a</sup>: Only for subjects requiring medication/therapy washout; X<sup>b</sup>: Re-draw blood and urine samples for clinical laboratory evaluations only if washout duration exceeded 5 weeks. <sup>C</sup> PK Schedule 1, PK Schedule 2, or PK Schedule 3 should be performed at selected sites based on what the subject chose in the ICF, <sup>d</sup>For subjects participating in PK Schedule 3 only.

#### <u>5.0</u> <u>OBJECTIVES</u>

The primary objective is to evaluate the efficacy of oral sarecycline 1.5 mg/kg/day compared to placebo in treating inflammatory acne lesions in subjects with moderate to severe facial acne vulgaris based on Investigator's Global Assessment score and inflammatory lesion counts.

The secondary objectives are to evaluate the safety of oral sarecycline 1.5 mg/kg/day based on adverse events, vital signs, electrocardiograms, physical examinations and clinical laboratory tests.

#### <u>6.0</u> <u>ANALYSIS POPULATIONS AND DATASETS</u>

#### 6.1 SCREENED POPULATION

The Screened Population will consist of all subjects who underwent a Screening Visit 1 and received a subject identification number (SID).

#### 6.2 SAFETY POPULATION

The Safety Population will consist of all subjects who received at least one dose of investigational product. All summaries of this population will be based on the treatment group each subject actually received.

#### 6.3 INTENT-TO-TREAT POPULATION

The Intent-to-Treat (ITT) Population will consist of all randomized subjects. All summaries of this population will be based on the treatment group each subject was randomized to receive.

#### 6.4 PER-PROTOCOL POPULATION

Per-protocol (PP) population will consist of all subjects in ITT population, as defined below. All summaries of this population will be based on the treatment group each subject was randomized to receive.

Subjects with the following conditions will be excluded from the PP population:

- 1. Did not meet inclusion/exclusion criteria
- 2. Have taken any interfering concomitant medications
- 3. Duration of treatment less than 68 days, or did not complete study based on subject exit status, or overall study drug compliance less than 80%
- 4. Received treatment different from the assigned treatment

A list of subjects with conditions 1, 2, and 3 above prior to unblinding will be created. This list will be reviewed by a Clinical Representative to determine which subjects are to be excluded from the PP population. These subjects will then be documented in a signed memo prior to unblinding. The subjects who received treatment different from the assigned treatment (condition 4) will be identified after unblinding and will be documented in a separate signed memo.

Three "visit types" will be defined for the purposes of analysis and summaries:

Observed Cases (OC) – includes assessments collected at each scheduled visit. All
applicable efficacy and safety variables will be summarized for OC visits.

- Multiple Imputation Data for the primary and secondary efficacy endpoints, missing data will be imputed using multiple imputation procedures further described in Section 16.2.
- LOCF defined as the last post-baseline data recorded for each efficacy variable.
   This visit will be denoted as Week 12 (LOCF) and will only be used to summarize efficacy data. The LOCF visit provides missing value imputation for subjects who do not provide data for the Week 12 visit.

#### 7.0 SUBJECT DISPOSITION

The number and percentage of subjects in 3 of the study populations (Safety, ITT and PP) will be summarized by treatment group and study center; the Screened Population will be summarized overall only by study center.

Screen-failure subjects (ie, subjects screened but not randomized) and the associated reasons for failure to randomize will be tabulated overall for the Screened Population. The number and percentage of subjects who complete the treatment period and of subjects who prematurely discontinue during the same period will be presented for each treatment group and pooled across treatment groups for the ITT Population. The reasons for premature discontinuation from the treatment period as recorded on the termination pages of the electronic case report forms (eCRF) will be summarized (number and percentage) by treatment group for the ITT Population. All subjects who prematurely discontinue during the treatment period will be listed by discontinuation reason for the ITT Population.

All subjects who are in ITT Population but not in PP Population will be listed with reasons provided.

# 8.0 DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS

Demographic parameters (age; age group ( $\geq$  9 years and < 18 years vs.  $\geq$  18 years); age group ( $\geq$  9 years and < 12 years,  $\geq$  12 years and < 18 years, and  $\geq$  18 years); race; sex; weight; weight group (33 to 54 kg, 55 to 84 kg, and 85 to 136 kg), height; body mass index (BMI), calculated as weight [kg]/(height [m])<sup>2</sup>; BMI group (< 25 kg/m<sup>2</sup> vs.  $\geq$  25 kg/m<sup>2</sup>); and hormonal contraceptive use in females) and other baseline characteristics (inflammatory lesion counts, IGA score, and IGA scores for neck, chest, and back sites) will be summarized descriptively by treatment group for the Safety, ITT, and PP populations. Weight rounding for weight group is in the following way: 54.4 to 54, 54.5 to 55. Continuous variables will be summarized by number of subjects and mean, median, SD, minimum, and maximum values. Categorical variables will be summarized by number and percentage of subjects.

Comparability between treatment groups for efficacy variables will be tested using a 2-way analysis-of-variance model with treatment group and study center as the factors for continuous variables (inflammatory lesion counts and IGA score) and the CMH test, controlling for study center, for the categorical variable of IGA score. Because of their clinical importance, IGA score of the baseline characteristics will be treated as both a continuous and categorical variable.

Abnormalities in subjects' medical and surgical histories will be coded using the *Medical Dictionary for Regulatory Activities*, version 18.0 or newer. The number and percentage of subjects with abnormalities in medical and surgical histories in each system organ class and preferred term will be summarized by treatment group and overall for the Safety Population.

Prior medications including acne medications are those medications with an end date before the date of the first dose of investigational product. Concomitant medications including acne medications are those medications with either 1) a start date that is after the first dose of investigational product, 2) a start date prior to the first dose of investigational product with end date on or after the date of first dose of investigational product, or 3) a start date prior to the first dose of investigational product and its use is ongoing. Any concomitant medications taken after the date of the last visit will not be presented in the summary tables but will be included in the subject data listings.

Both prior and concomitant medications will be coded by drug preferred name and therapeutic class. The use of prior and concomitant medications and the use of prior and concomitant acne medications will be summarized by the number and percentage of subjects in each treatment group and overall for the Safety Population. If a subject took a specific medication multiple times or took multiple medications within a specific therapeutic class, that subject would be counted only once for the coded drug preferred name or therapeutic class.

The World Health Organization (WHO) Drug Dictionary, version March 2015 or newer, will be used to classify prior and concomitant medications by WHO Drug Anatomical/Therapeutic/Chemical category and WHO Drug preferred name.

#### 9.0 EXTENT OF EXPOSURE AND TREATMENT COMPLIANCE

#### 9.1 EXTENT OF EXPOSURE

Exposure to the investigational product for the Safety Population during the double-blind treatment period will be summarized for treatment duration, calculated as the number of days from the date of the first dose of the investigational product to the date of the last dose of the double-blind investigational product, inclusive. Descriptive statistics (number of subjects, mean, SD, median, minimum, and maximum) will be presented by treatment group. Additionally, these summaries will present the number and percentage of subjects for each interval (1 week multiples) of total exposure in each treatment. The denominators for calculating the percentages will be based on the number of subjects with exposure for each treatment.

Subjects in the PK Schedule 3 group who receive one active dose of study drug after study assessments at Week 12 will also be listed (separately) for this single-dose exposure.

#### 9.2 MEASUREMENT OF TREATMENT COMPLIANCE

Dosing compliance for a specified period is defined as the number of tablets actually taken by a subject during that period divided by the expected number of tablets taken for the same period multiplied by 100. This information will be obtained from the drug accountability of the subject's eCRF. The total number of tablets actually taken will consist of subtracting both the total numbers of tablets returned and the total numbers of tablets lost from the total number of tablets dispensed. The number of tablets expected to be taken for a specific treatment period will be calculated based on the number of days in that period. Descriptive statistics for dosing compliance will be presented by treatment group for the whole double-blind treatment period for the Safety Population.

#### <u>10.0</u> <u>EFFICACY ANALYSES</u>

The efficacy analyses will be based on the ITT Population. All summaries on this population will be based on the investigational product each subject was randomized to receive. The multiple imputation (MI) approach will be used to impute missing values for co-primary and secondary efficacy analyses and details are further described in Section 16.2. Sensitivity analyses for efficacy parameters will be performed using alternative approaches to handle missing data, as well as an observed cases (OC) approach using the PP population. *Baseline* for efficacy is defined as the last non-missing efficacy assessment before the first dose of the investigational product. All statistical tests will be 2-sided hypothesis tests performed at the 5% level of significance for main effects. All confidence intervals will be 2-sided 95% confidence intervals, unless stated otherwise.

The descriptive statistics for all the continuous variables will include the mean, median, 25th percentile, 75th percentile, standard deviation (SD), standard error of mean (SEM), minimum, maximum, and number of subjects. Descriptive summaries will be provided for raw, change from baseline (CFB), and %CFB values for continuous efficacy endpoints. Frequency distributions for all the categorical variables will be presented as counts and percentages. Summaries will be provided by visit and treatment, as appropriate.

While every effort will be made to randomize a sufficient number of subjects at each study site, in the event that this is not possible, study sites may be pooled for statistical inference testing. Study sites (centers) will be pooled by geographical location based on region definitions from the US Census Bureau (Northeast, Midwest, South, and West; US Census Bureau, 2013) for analysis purposes so that in each pooled site the number of subjects is reasonably large and consistent in size between pooled sites. Sites within a geographic location will be pooled starting with the sites that have the lowest number of randomized subjects pooled together such that the pooled site has a minimum of 12 randomized subjects after pooling.

The sites to be pooled for each geographic location will be documented in a signed memo prior to unblinding of the treatment code. A list of sites and the corresponding pooled sites will be presented.

#### 10.1 CO-PRIMARY EFFICACY PARAMETERS

There will be two co-primary efficacy parameters (endpoints) for this study. The first coprimary efficacy endpoint will be the absolute CFB in inflammatory lesion counts at Week 12. This variable will be considered a continuous variable. The second co-primary efficacy endpoint will be IGA success at Week 12. IGA success will be a dichotomous variable defined as at least 2-point decrease from baseline on the IGA assessment as well as a score of clear (0) or almost clear (1) on the IGA assessment.

#### 10.1.1 CFB in Inflammatory Lesion Counts

The co-primary endpoint, absolute CFB in inflammatory lesion counts at Week 12, will be analyzed using an analysis of covariance (ANCOVA) model with the baseline value as a covariate and additional terms included to represent effects of treatment and (pooled) site. The primary efficacy analysis will be based on the ITT population. Missing data will be imputed using an MI approach further described in Section 16.2. The adjusted means with associated 95% confidence intervals (CIs) from the ANCOVA model will also be presented for each treatment and for the difference between the treatments. Statistical significance between the treatments, sarecycline compared to placebo, will be declared if the p-value of the hypothesis test from the ANCOVA model is less than or equal to 0.05. The ANCOVA model will be performed using SAS® PROC MIXED with the methodology of Littell et al. (2006).

Let  $X_{ijk}$  and  $Y_{ijk}$  be the baseline and endpoint values for the kth subject in the jth site and the ith treatment, where  $k=1,...,n_j$ , j=1,...,c (the number of sites after pooling, if applicable) and i=sarecycline, placebo. Then

$$Y_{ijk} - X_{ijk} = \mu + \tau_i + \gamma_j + \beta X_{ijk} + \varepsilon_{ijk}$$

where  $\mu$  is the overall mean,  $\tau$  is the fixed effect of the *i*th treatment,  $\gamma$  is the fixed effect of the *j*th site,  $\beta$  is a regression coefficient for baseline and  $\epsilon_{ijk}$  is the NID(0, $\sigma^2$ ) random error component. Hypothesis tests for the active treatment effect of sarecycline compared to placebo will be conducted using differences of adjusted means.

As site is included in the primary ANCOVA model, a treatment-by-site interaction will be investigated as an exploratory analysis to assess the homogeneity of treatment effects across site. This effect will be investigated analytically prior to any pooling of sites by adding the interaction term to the ANCOVA model and testing for significance. Because interactions are not powered in this study, testing for significance will be at the 0.10 level. However, any significant interaction findings at the 0.10 level will also take into account the potential for spurious results. Further exploration may be done graphically with interaction plots to determine the nature of the interaction and to identify any "outlier" sites with attention focused on qualitative differences in treatment effects. If large differences in treatment effects are seen in any "extreme" sites, then sensitivity analyses will be performed that exclude sites with the highest extreme treatment effect values from the analysis. Any such sites may be further investigated for explanation involving study conduct, subject demographics, current medications, etc.

In addition, the following sensitivity analyses will be performed:

 Inflammatory lesion count data will be analyzed for CFB at Week 12 according to an ANCOVA model with the baseline value as a covariate and effects of treatment and (pooled) site using the PP population with OC data.

- LOCF will be used as an imputation method for cases where the Week 12 CFB in
  inflammatory lesion counts value is missing. The endpoint will then be analyzed
  according to an ANCOVA model with the baseline value as a covariate and effects of
  treatment and (pooled) site.
- Baseline observation carried forward will be used as an imputation method for cases
  where the Week 12 CFB in inflammatory lesion counts value is missing. The
  endpoint will then be analyzed according to an ANCOVA model with the baseline
  value as a covariate and effects of treatment and (pooled) site.
- Mixed model repeated measures (MMRM) analysis will be used to explore the sensitivity of data handling for CFB in inflammatory lesion counts for subjects who withdraw from the study. The model will include the fixed effects of treatment, pooled site, and visit, the baseline value as a covariate, and the treatment-by-visit interaction term. An unstructured covariance matrix will be used initially in the model for the correlation pattern among the repeated measures. If this does not converge, then the Toeplitz covariance structure (TYPE=TOEP in SAS MIXED procedure) will be used instead. If the results from the MMRM analyses differ qualitatively with the results from the primary efficacy analysis, further analyses will be performed to investigate the causes of the difference. However, the results from the primary efficacy analysis will be considered the primary efficacy results.
- A rank transformation will be applied to each of the multiple datasets created from the MI approach and the analysis will proceed for Week 12 using an ANCOVA model on the ranks with the baseline value as a covariate and effects of treatment and (pooled) site. Tied values will receive the mean value (midranks) of the corresponding ranks.

#### 10.1.2 IGA Success

The co-primary efficacy endpoint, percentage of subjects with IGA success at Week 12, will be analyzed for the ITT population using the CMH test with adjustment for (pooled) site. Missing data will be imputed using an MI approach further described in Section 16.2. The rate difference and the 95% CIs for the rate difference and the relative rate and the 95% CIs for the relative rate will be presented as well. The CI for the treatment rate difference will be based on two-sided 95% Wald type CIs with CMH weights (Kim & Won, 2013, Yan & Su, 2010).

The homogeneity of treatment effects across (pooled) site will be investigated as an exploratory analysis using the Breslow-Day test. If the Breslow-Day test indicates large heterogeneity in the odds ratios across (pooled) site, then further exploration may be done graphically or with further investigation for explanation involving study conduct, subject demographics, current medications, etc.

In addition, the following sensitivity analyses will be performed:

- IGA success at Week 12 will be analyzed using a CMH test with adjustment for (pooled) site on the PP population with OC data.
- For IGA success, subjects who discontinue from the study early will be coded as
  failures for the Week 12 analysis. A sensitivity analysis of IGA success using this
  data handling convention will be performed using a CMH test with adjustment for
  (pooled) site.
- For IGA success, subjects who discontinue from the study early will be coded as
  failures for subjects on sarecycline and successes for subjects on placebo. A
  sensitivity analysis of IGA success using this data handling convention will be
  performed using a CMH test with adjustment for (pooled) site.

#### 10.2 SECONDARY EFFICACY PARAMETERS

There will be 8 sets of secondary efficacy endpoints for this study: percent CFB in inflammatory lesion counts at Week 12, absolute and percent CFB in inflammatory lesion counts at Weeks 9, 6, and 3, and absolute and percent CFB in noninflammatory lesion counts at Weeks 12, 9, 6, and 3. These variables will be considered continuous variables.

A hierarchical testing approach will be used for the secondary efficacy endpoints, such that statistical testing will only be performed if both co-primary efficacy endpoints are statistically superior to placebo at  $\alpha$ =0.05. In addition, statistical testing of the secondary endpoints will be conducted in the following order, with all tests proceeding at the 0.05 level if and only if the previous tests were all significant at the 0.05 level:

- 1. Percent CFB for inflammatory lesion counts at Week 12
- 2. Absolute and percent CFB for inflammatory lesion counts at Week 9 (both endpoints must be significant at the 0.05 level to proceed to the next analyses)
- 3. Absolute and percent CFB for inflammatory lesion counts at Week 6 (both endpoints must be significant at the 0.05 level to proceed to the next analyses)
- 4. Absolute and percent CFB for inflammatory lesion counts at Week 3 (both endpoints must meet the 0.05 level for Week 3 to meet statistical significance)
- 5. Absolute and percent CFB for noninflammatory lesion counts at Week 12 (both endpoints must be significant at the 0.05 level to proceed to the next analyses)
- 6. Absolute and percent CFB for noninflammatory lesion counts at Week 9 (both endpoints must be significant at the 0.05 level to proceed to the next analyses)
- 7. Absolute and percent CFB for noninflammatory lesion counts at Week 6 (both endpoints must be significant at the 0.05 level to proceed to the next analyses)

8. Absolute and percent CFB for noninflammatory lesion counts at Week 3 (both endpoints must meet the 0.05 level for Week 3 to meet statistical significance)

These endpoints will be analyzed for each visit using an analysis of covariance (ANCOVA) model with terms included to represent effects of treatment and (pooled) site and the baseline values as a covariate for the ITT population. Missing data will be imputed using an MI approach, as described in Appendix 16.2. The adjusted means with associated 95% CIs for the ANCOVA model will also be presented for each treatment and for the difference between the treatments. Statistical significance between the treatments, sarecycline compared to placebo, will be declared if the p-value of the hypothesis test from the ANCOVA model is less than or equal to 0.05.

For the Week 12 percent CFB analysis, as site is included in the ANCOVA model, a treatment-by-site interaction will be investigated as an exploratory analysis to assess the homogeneity of treatment effects across site. This effect will be investigated analytically by adding the interaction term to the ANCOVA model and testing for significance. Because interactions are not powered in this study, testing for significance will be at the 0.10 level. However, any significant interaction findings at the 0.10 level will also take into account the potential for spurious results with attention focused on qualitative differences in treatment effects. If large differences in treatment effects are seen in any "extreme" sites, then sensitivity analyses will be performed that exclude sites with the highest extreme treatment effect values from the analysis. Further exploration may be done graphically with interaction plots to determine the nature of the interaction and to identify any "outlier" sites. Any such sites may be further investigated for explanation involving study conduct, subject demographics, current medications, etc.

An additional exploratory analysis will be done for the percent CFB analysis by visit. A rank transformation will be applied to each of the multiple datasets created from the MI approach and the analysis will proceed using an ANCOVA model on the ranks with the baseline value as a covariate and effects of treatment and (pooled) site. Tied values will receive the mean value (midranks) of the corresponding ranks.

# 10.3 ADDITIONAL EFFICACY PARAMETER



#### 10.4 SUBGROUP ANALYSES

Primary and secondary efficacy variable summaries will be repeated for the following subgroups by study visit using OC data:

- · Gender: male and female
- Age groups: >= 9 and < 18 years; ≥ 18 years</li>
- Race: white, African-American/Black, other
- Body mass index:  $< 25 \text{ kg/m}^2 \text{ and } \ge 25 \text{ kg/m}^2$
- Baseline acne severity (IGA score): moderate and severe
- Hormonal contraceptive use in females: female subjects who use hormonal contraceptives versus female subjects who do not
- Weight groups: 33 to 54 kg, 55 to 84 kg, and 85 to 136 kg

#### 10.5 OTHER EFFICACY PARAMETERS

#### 10.5.1 IGA for Non-facial Sites



#### 10.5.2 Skindex Questionnaire

| | | | | _ |
|------|-------------------|-----------|----|---|
| 10.6 | ADDITIONAL EFFICA | CY ANALYS | ES | |

#### 11.0 SAFETY ANALYSES

The safety analysis will be performed using the Safety Population. The safety parameters will include adverse events (AEs) and clinical laboratory, vital sign, ECG, and noninflammatory lesion counts parameters. For each safety parameter of the clinical laboratory, vital sign, ECG parameters, and noninflammatory lesion counts parameters, the last nonmissing safety assessment on or before the date of the first dose of the investigational product will be used as the baseline for all analyses of that safety parameter. Continuous variables will be summarized by number of subjects and mean, SD, median, minimum, and maximum values. Categorical variables will be summarized by number and percentage of subjects.

#### 11.1 ADVERSE EVENTS

Adverse events will be coded by system organ class and preferred term using the *Medical Dictionary for Regulatory Activities*, version 18.0 or newer.

Adverse events with onset on or after the first dose date of the study drug will be considered as "treatment-emergent adverse event (TEAE)". An AE that occurs more than 30 days after the date of the last dose of the investigational product will not be counted as a TEAE. Adverse events summaries will present the number and percentage of subjects reporting an adverse event by treatment and overall as well as the number of events reported. The denominators for calculating the percentages by treatment will be based on the number of subjects exposed in the Safety population to each treatment and overall. The treatment will be based on the double-blind treatment received. For subjects who are in PK schedule 3, the TEAE summary described will comprise data prior to the active dose taken at the Week 12 visit. Further adverse events experienced after this Week 12 dose will be listed separately for these subjects.

The number and percentage of subjects reporting TEAEs in each treatment group and overall will be tabulated by system organ class and preferred term and further categorized by severity and relationship to study treatment. If more than 1 AE is coded to the same preferred term for the same subject, the subject will be counted only once for that preferred term using the greatest severity and strictest causality for the summarization by severity and relationship.

The incidence of common ( $\geq 2\%$  of subjects in any treatment group) TEAEs will be summarized by preferred term and treatment group and will be sorted by decreasing frequency for sarecycline treatment group.

The total number of TEAEs by severity and relationship to study treatment will be summarized by treatment group.

A serious adverse event (SAE) that occurred between the date of the first dose of the investigational product and 30 days after the date of the last dose of the investigational product, inclusive, will be considered an on double-blind therapy SAE. However, for any subject in the PK schedule 3 group, SAEs that occur after the Week 12 active dose will not be included. These events will be listed separately. The number and percentage of subjects who have on-therapy SAEs will be summarized by preferred term and treatment group and will be sorted by decreasing frequency for sarecycline treatment group. In addition, the incidence of on-therapy SAEs that led to death will be summarized separately by preferred term for each treatment group.

The number and percentage of subjects in the Safety Population who have AEs leading to premature discontinuation of the investigational product will be summarized by preferred term and treatment group and will be sorted by decreasing frequency for sarecycline treatment group.

Gastrointestinal AEs of special interest will be pre-specified prior to database lock. The number and percentage of subjects in the Safety Population who have gastrointestinal TEAEs of special interest will be summarized by preferred term and treatment group and will be sorted by decreasing frequency for sarecycline treatment group. In addition, these TEAEs will be further categorized by relationship to study treatment.

For the Screened Population, separate tabular displays will be presented for subjects who died, subjects with SAEs, and subjects with AEs leading to premature discontinuation.

#### 11.2 CLINICAL LABORATORY PARAMETERS

Descriptive statistics for clinical laboratory values (in SI units) and changes from the baseline values at each assessment time point will be presented by double-blind treatment group for the following laboratory analytes:

Hematology: Hemoglobin, hematocrit, red blood cell count, mean cell volume,

white blood cell count, white blood cell count differential, and platelet

count

Chemistry: albumin, alanine aminotransferase, aspartate aminotransferase, blood

urea nitrogen, gamma glutamyl transferase, glucose, lactate,

dehydrogenase, total bilirubin, creatine phosphokinase, total protein, serum creatinine, sodium potassium, calcium, chloride, bicarbonate,

and phosphorus

Urinalysis: color, specific gravity, potential for hydrogen (pH), leukocytes,

ketones, protein, glucose, blood, and bilirubin

Lipid Profile: total cholesterol and triglycerides

Thyroid Function: thyroid stimulating hormone and free T4 and T3

#### Other Urine pregnancy test

Continuous clinical laboratory analytes will be summarized by double-blind treatment, analyte, and visit using descriptive statistics. Categorical laboratory analytes, classified as normal or abnormal (low or high), will be summarized by double-blind treatment group,

Clinical laboratory test values will be considered potentially clinically significant (PCS) if they meet either the lower-limit or higher-limit criteria provided by the (Appendix 1). The number and percentage of subjects who have PCS postbaseline clinical laboratory values will be tabulated by double-blind treatment group for the treatment period. The percentages will be calculated relative to the number of subjects with available non-PCS baseline values and at least 1 postbaseline assessment for the treatment period. The numerator will be the total number of subjects with available non-PCS baseline values and at least 1 PCS postbaseline value for the treatment period. A supportive tabular display of subjects with PCS postbaseline values will be provided, including SID, study center number, and baseline and all postbaseline (including non-PCS) values.

In addition, a tabular display showing all AEs that occurred in subjects who had PCS postbaseline clinical laboratory values will be provided.

Shift tables from baseline to end of the double-blind study period for clinical laboratory parameters will be presented by treatment group for the following categories: low, normal, and high.

Subjects with potential drug induced liver injury (elevated AST or ALT 3 times upper limit of normal (ULN) or greater and elevated bilirubin greater than 2 times ULN) will be listed. In addition, a tabular display showing all AEs that occurred in subjects with potential drug induced liver injury will be provided.

#### 11.3 VITAL SIGNS

Descriptive statistics for vital signs (systolic and diastolic blood pressures, heart rate, and weight) and changes from baseline values at each visit and at the end of the double-blind study period will be presented by treatment group.

Vital sign values will be considered PCS if they meet both the observed-value criteria and the change-from-baseline criteria listed in Table 11.3–1. The number and percentage of subjects with PCS postbaseline values will be tabulated by treatment group for the double-blind treatment period. The percentages will be calculated relative to the number of subjects with available baseline values and at least 1 postbaseline assessment for the treatment period. The numerator will be the total number of subjects with available baseline values and at least 1 PCS postbaseline value for the treatment period. A supportive tabular display of subjects with PCS postbaseline values will be provided, including SID, study center number, and baseline and all postbaseline (including non-PCS) values.

In addition, a tabular display showing all AEs that occurred in subjects who had PCS postbaseline vital sign values will be provided.

Shift tables from baseline to end of the double-blind study period for vital signs (systolic and diastolic blood pressures, pulse rate) will be presented by treatment group for the following categories: low, normal, and high

Table 11.3–1. Criteria for Potentially Clinically Significant Vital Signs

| Vital Sign | Age | Gender | Flag | Criterion Value |
|---|---|---|---|---|
| Systolic blood pressure, mm Hg | 9 to 45 | Female or<br>Male | High | > 140 |
| Diastolic blood pressure, mm Hg | 9 to 45 | Female of<br>Male | High | ≥ 90 |
| | 9 to 12 | Female | High | > 121 |
| | | | Low | < 50 |
| | 9 to 12 | Male | High | > 112 |
| | | | Low | < 49 |
| | 13 to 16 | Female | High | > 118 |
| Heart rate, beats per minute | | | Low | < 48 |
| | 13 to 16 | Male | High | > 110 |
| | | | Low | < 42 |
| | 17 to 45 | Female or<br>Male | High | > 110 |
| | 17 to 45 | Female or<br>Male | Low | < 44 |

#### 11.4 ELECTROCARDIOGRAM

Descriptive statistics for ECG parameters (heart rate, RR interval, PR interval, QRS duration, QT interval, and QTc) and changes from baseline values at each assessment time point to the end of the double-blind study period will be presented by treatment group. The QTc will be calculated using both the Bazett and Fridericia corrections.

Electrocardiographic parameter values are considered PCS if they meet or exceed the higher-limit PCS criteria listed in Table 11.4–1. The number and percentage of subjects with PCS postbaseline ECG values will be tabulated by treatment group for the double-blind treatment period. The percentages will be calculated relative to the number of subjects with available non-PCS baseline values and at least 1 postbaseline assessment for the treatment period. The numerator is the total number of subjects with available non-PCS baseline values and at least 1 PCS postbaseline value for the treatment period. A supportive tabular display of subjects with PCS postbaseline values will be provided, including SID, study center number, baseline, all postbaseline (including non-PCS) values, and change from baseline.

In addition, a tabular display showing all AEs that occurred in subjects who had postbaseline PCS ECG values will be provided.

A shift table from baseline to the end of the double-blind study in the Investigator's overall interpretation of the ECG will be presented by treatment group for the following categories: normal; abnormal, not clinically significant; abnormal, clinically significant. A tabular display showing subjects with postbaseline clinically significant ECG abnormalities according to the Investigator's overall interpretation will be provided.

Table 11.4–1. Criteria for Potentially Clinically Significant Electrocardiograms

| Parameter | Unit | Higher Limit |
|-----------------------------|------|----------------|
| QRS duration | msec | ≥ 120 |
| PR interval | msec | > 220 or < 110 |
| QTc (QTcB or QTcF) interval | msec | > 500 |

QTc = QT interval corrected for heart rate.

#### 11.5 OTHER SAFETY PARAMETERS

#### 11.5.1 Noninflammatory Lesion Counts

Noninflammatory lesions (open and closed comedones) will be counted and recorded in the eCRF and will be analyzed for CFB using an ANCOVA model effects of treatment, (pooled) site, and the baseline value as a covariate using OC data. Note that non-inflammatory lesion counts serve as both a safety and efficacy parameter in this study, reflecting a dual role of assessing efficacy while also evaluating patient safety.

## 12.0 HEALTH OUTCOMES ANALYSES

No health outcome analyses are planned for this study.

## 13.0 INTERIM ANALYSIS

No interim analysis is planned for this study.

#### <u>14.0</u> <u>DETERMINATION OF SAMPLE SIZE</u>

The sample size was selected to provide an adequate number of subjects to compare the efficacy of sarecycline treatment to placebo and to provide an adequate number of subjects needed for a safety database.

Sample size estimates were calculated for each of the co-primary efficacy endpoints, absolute CFB in facial inflammatory lesion counts and facial IGA success (based on at least 2-point decrease from baseline in IGA score), and the first secondary efficacy endpoint, percent CFB in facial inflammatory lesion counts at Week 12 last observation carried forward (LOCF). The results from a recent study (Study PR-10411) of sarecycline compared to placebo treatment were used to estimate the sample size needed to show a significant difference between the treatments at  $\alpha$ =0.05 and 90% power using two-sided tests and a 1:1 randomization. It should be noted that one outlier in the data for Study PR-10411 was removed from the estimate for absolute CFB in inflammatory lesion counts in order to provide more accurate estimates for the sample size determination. Results of the calculations and the estimates used in the calculations are provided below:

| Continuous<br>Endpoints <sup>a</sup> | Sarecycline<br>CFB or %CFB | Placebo<br>CFB or %CFB | Common<br>SD | Sample per<br>Treatment | Total<br>Sample Size |
|---|---|---|---|---|---|
| Absolute CFB in inflammatory lesion counts (co-primary) | 16 | 13 | 12 | 338 | 676 |
| Percent CFB in<br>inflammatory lesion<br>counts (secondary) | 52% | 39% | 41% | 210 | 420 |

a Sample size was based on a two sample t-test of no difference between the treatments

| Dichotomous | Sarecycline | Placebo | Difference in | Sample per | Total |
|---|---|---|---|---|---|
| Endpoints <sup>a</sup> | Rate | Rate | Rates | Treatment | Sample Size |
| IGA Success<br>(2-point decrease in IGA<br>score from baseline and a<br>score of clear/almost clear;<br>co-primary) | 23% | 10% | 13% | 170 | 340 |

a Sample size was based on a  $\chi^2$  test of no difference between the proportions

While the IGA scale proposed for the Phase 2 study is slightly different than the IGA scale in the Phase 2, the number of subjects to be enrolled (500 per treatment; 1000 total) should provide more than sufficient power for the efficacy evaluations. Additionally, a larger sample is needed in order to provide sufficient numbers of subjects on sarecycline treatment for a safety database.

## 15.0 STATISTICAL SOFTWARE

Statistical analyses will be performed using version 9.3 (or newer) of SAS on a LINUX operating system.

#### <u>16.0</u> <u>DATA HANDLING CONVENTIONS</u>

#### 16.1 VISIT TIME WINDOWS

Table 16.1–1 presents the visits assigned for efficacy and safety analyses and the corresponding range of treatment days (window) during which an actual visit may occur.

Table 16.1–1. Visit Time Windows

| Derived Visit | Scheduled Visit Day <sup>a</sup> | Window |
|---|---|---|
| Baseline | Day 1 | Days ≤ 1 |
| Week 3 | Day 22 | Days [2, 32] |
| Week 6 | Day 43 | Days [33, 53] |
| Week 9 | Day 64 | Days [54, 74] |
| Week 12 | Day 85 | Days ≥ 75 |
| End of study <sup>b</sup> | Final or Termination Visit during the treatment period | |

a Relative to the date of the first dose of the investigational product or date of randomization if patient did not receive any dose. Day 1 = the date of the first dose of the investigational product (or date of randomization if patient did not receive a dose). There is no Day 0.

If the assessment date ( if the assessment date is unavailable, using visit date instead) is on or after the date of the first dose of the investigational product, the study day is calculated by assessment date – date of the first dose of the investigational product + 1. If the assessment date is before the date of the first dose of the investigational product, the study day is calculated by assessment date – date of the first dose of the investigational product. Therefore, a negative day indicates a day before the start of the investigational product.

If a subject has 2 or more visits within the same window, the last visit with a nonmissing value will be used for analysis.

# 16.2 MISSING DATA HANDLING FOR PRIMARY AND SECONDARY EFFICACY ENDPOINTS

For the co-primary and secondary efficacy analyses, the primary missing data imputation method is multiple imputation, as outlined in the following procedures:

The SAS PROC MI procedure with a fully conditional specifications (FCS) method will be used to create 20 imputations. The FCS is proposed as it allows for accommodation of categorical variables and it has the versatility to handle arbitrary missing data patterns. Based on these 20 imputations, the relative efficiency will be 0.995 for 10% of missing data and 0.990 for 20% of missing data (Rubin, 1976, 1987, 1996).

b Presented in analysis tables for safety parameters, including but not limited to electrocardiograms, clinical laboratory values, and vital signs.

- o For inflammatory lesion counts, if any of the subtypes (papules, pustules, and nodules/cysts) is missing, the inflammatory lesion count is missing. The variables included in the imputations are age, gender, and the measurements of the corresponding endpoint count) at baseline, Week 3, Week 6, Week 9, and Week 12.
- For IGA, the raw scores will be used for the imputation. The variables included in the imputations are age, gender, and the measurements of the endpoint at baseline, Week 3, Week 6, Week 9, and Week 12.
- All imputations will be performed by treatment group based on the randomized study medication and based on the randomized gender strata. The number of imputation is set at 20 with number of 50 burn-in iterations. The seed used for imputation for all endpoints is \_\_\_\_\_\_. The logistic regression model for gender is based on the probability of female. For age, IGA raw scores and lesion counts, regression with predictive mean matching method will be used. The imputed values will be rounded to the nearest integer for IGA and lesion counts.
- The following are the SAS programs used to impute IGA at week 12:



The following SAS program will be used to impute inflammatory and non-inflammatory lesion counts at week 12.



- An analysis of covariance (ANCOVA) model for inflammatory lesion counts and a CMH analysis for the IGA success as stated in Sections 10.1.1 and 10.1.2, respectively, will be performed for each of the imputed dataset.
- An analysis of covariance (ANCOVA) model for inflammatory and noninflammatory lesion counts as stated in Section 10.2 will be performed for the imputed dataset for the secondary endpoints.
- The SAS PROC MIANALYZE procedure will be used to produce final parameter estimates, including the point estimates and standard errors, adjusted treatment differences, confidence intervals and p-values for the primary and secondary variables.
- For the CMH test, the Wilson-Hilferty transformation (Wilson & Hilferty, 1931, O'Kelly & Ratitch, 2014) will be used. Under the null hypothesis, the transformed statistic is approximately normally distributed:

$$wh\_CMH^{(m)} = \sqrt[3]{\frac{cmh^{(m)}}{k}} \sim normal(1 - \frac{2}{9k}, \frac{2}{9k})$$

Where  $cmh^{(m)}$  is the chi-square statistics each with k degrees of freedom from m = 1, ..., M imputed datasets. In this case, k=1. This statistic will be passed to PROC MIANALYZE to obtain the combined p-value for CMH test.

The same method will be used to obtained the p-values from the Breslow-Day test.

# 16.3 REPEATED OR UNSCHEDULED ASSESSMENTS OF SAFETY PARAMETERS

If a subject has repeated assessments before the start of investigational product, the results from the final nonmissing assessment made before the start of the investigational product will be used as baseline. If end-of-study assessments are repeated or if unscheduled visits occur, the last nonmissing postbaseline assessment will be used as the end-of-study assessment for generating summary statistics. However, all postbaseline assessments will be used for PCS value determinations, and all assessments will be presented in the data listings.

## 16.4 MISSING DATE OF THE LAST DOSE OF INVESTIGATIONAL PRODUCT

When the date of the last dose of the investigational product is missing for a subject in the Safety Population, all efforts should be made to obtain the date from the Investigator. If after all efforts are made it is still missing, the last available dosing record date will be used as the last dose date.

#### 16.5 MISSING SEVERITY ASSESSMENT FOR ADVERSE EVENTS

If severity is missing for an AE that started before the date of the first dose of the investigational product, an intensity of mild will be assigned. If severity is missing for an AE that started on or after the date of the first dose of the investigational product, an intensity of severe will be assigned. The imputed values for severity assessment will be used for the incidence summary; the values will be shown as missing in the data listings.

# 16.6 MISSING RELATIONSHIP TO INVESTIGATIONAL PRODUCT FOR ADVERSE EVENTS

If the relationship to study treatment is missing for an AE that started on or after the date of the first dose of the investigational product, a relationship of related will be assigned. The imputed values for relationship to study treatment will be used for the incidence summary; the values will be shown as missing in the data listings.

#### 16.7 MISSING DATE INFORMATION FOR ADVERSE EVENTS

The following imputation rules only apply to cases in which the start date for AEs is incomplete (ie, partly missing).

#### Missing month and day

- If the year of the incomplete start date is the same as the year of the first dose of the investigational product, the month and day of the first dose of the investigational product will be assigned to the missing fields
- If the year of the incomplete start date is before the year of the first dose of the investigational product, *December 31* will be assigned to the missing fields
- If the year of the incomplete start date is after the year of the first dose of the investigational product, *January 1* will be assigned to the missing fields

#### Missing month only

 If only the month is missing, the day will be treated as missing and both the month and the day will be replaced according to the above procedure
#### Missing day only

- If the month and year of the incomplete start date are the same as the month and year of the first dose of the investigational product, the day of the first dose of the investigational product will be assigned to the missing day
- If either the year of the incomplete start date is before the year of the date of the first
  dose of the investigational product or if both years are the same but the month of the
  incomplete start date is before the month of the date of the first dose of the
  investigational product, the last day of the month will be assigned to the missing day
- If either the year of the incomplete start date is after the year of the date of the first dose of the investigational product or if both years are the same but the month of the incomplete start date is after the month of the date of the first dose of the investigational product, the first day of the month will be assigned to the missing day

If the stop date is complete and the imputed start date as above is after the stop date, the start date will be imputed by the stop date.

If the start date is completely missing and the stop date is complete, the following algorithm will be used to impute the start date:

- If the stop date is after the date of the first dose of the investigational product, the date
  of the first dose of the investigational product will be assigned to the missing start
  date
- If the stop date is before the date of the first dose of the investigational product, the stop date will be assigned to the missing start date

## 16.8 MISSING DATE INFORMATION FOR PRIOR OR CONCOMITANT MEDICATIONS

For prior or concomitant medications, including rescue medications, incomplete (ie, partly missing) start dates and/or stop dates will be imputed. When the start date and the stop date are both incomplete for a subject, the start date will be imputed first.

#### 16.8.1 Incomplete Start Date

The following rules will be applied to impute the missing numeric fields for an incomplete prior or concomitant medication start date. If the stop date is complete (or imputed) and the imputed start date is after the stop date, the start date will be imputed using the stop date.

#### Missing month and day

If the year of the incomplete start date is the same as the year of the first dose of the
investigational product, the month and day of the first dose of the investigational
product will be assigned to the missing fields

- If the year of the incomplete start date is before the year of the first dose of the investigational product, *December 31* will be assigned to the missing fields
- If the year of the incomplete start date is after the year of the first dose of the investigational product, *January 1* will be assigned to the missing fields

#### Missing month only

• If only the month is missing, the day will be treated as missing and both the month and the day will be replaced according to the above procedure

#### Missing day only

- If the month and year of the incomplete start date are the same as the month and year of the first dose of the investigational product, the day of the first dose of the investigational product will be assigned to the missing day
- If either the year of the incomplete start date is before the year of the date of the first dose of the investigational product or if both years are the same but the month of the incomplete start date is before the month of the date of the first dose of the investigational product, the last day of the month will be assigned to the missing day.
- If either the year of the incomplete start date is after the year of the date of the first dose of the investigational product or if both years are the same but the month of the incomplete start date is after the month of the date of the first dose of the investigational product, the first day of the month will be assigned to the missing day

#### 16.8.2 Incomplete Stop Date

The following rules will be applied to impute the missing numeric fields for an incomplete prior or concomitant medication stop date. If the date of the last dose of the investigational product is missing, replace it with the last visit date in the imputations described below. If the imputed stop date is before the start date (imputed or nonimputed start date), the imputed stop date will be equal to the start date.

#### Missing month and day

- If the year of the incomplete stop date is the same as the year of the last dose of the investigational product, the month and day of the last dose of the investigational product will be assigned to the missing fields
- If the year of the incomplete stop date is before the year of the last dose of the investigational product, *December 31* will be assigned to the missing fields
- If the year of the incomplete stop date is after the year of the last dose of the investigational product, *January 1* will be assigned to the missing fields

#### Missing month only

• If only the month is missing, the day will be treated as missing and both the month and the day will be replaced according to the above procedure

#### Missing day only

- If the month and year of the incomplete stop date are the same as the month and year
  of the last dose of the investigational product, the day of the last dose of the
  investigational product will be assigned to the missing day
- If either the year of the incomplete stop date is before the year of the date of the last dose of the investigational product or if both years are the same but the month of the incomplete stop date is before the month of the date of the last dose of the investigational product, the last day of the month will be assigned to the missing day
- If either the year of the incomplete stop date is after the year of the date of the last dose of the investigational product or if both years are the same but the month of the incomplete stop date is after the month of the date of the last dose of the investigational product, the first day of the month will be assigned to the missing day

## 16.9 CHARACTER VALUES OF CLINICAL LABORATORY PARAMETERS

If the reported value of a clinical laboratory parameter cannot be used in a statistical summary table because, for example, a character string is reported for a parameter of the numeric type, a coded value must be appropriately determined for use in the statistical analyses. The actual values, however, as reported in the database will be presented in the data listings.

Table 16.9–1 shows examples of how some possible laboratory results should be coded for the analysis.

Table 16.9–1. Examples of Coding Special Character Values for Clinical Laboratory Parameters

| Laboratory Test,<br>SI Unit | Possible Laboratory Results | Coded Value for Analysis |
|---|---|---|
| CHEMISTRY | | |
| ALT, U/L | < 5 | 0 |
| AST, U/L | < 5 | 0 |
| Bilirubin, total, μmol/L | < 2 | 0 |
| URINALYSIS | | |
| Clusaca mmal/I | $= OR > 55, \ge 55, > 0$ | Positive |
| Glucose, mmol/L | $\leq$ 0, negative | Negative |
| »H | > 8.0, ≥ 8.0 | 8.0 |
| pH | ≥ 8.5 | 8.5 |
| Dustain | $= OR > 3.0, \ge 3.0, > 0$ | Positive |
| Protein | ≤0 | Negative |

 $\label{eq:all-linear} ALT = alanine aminotransferase; \ AST = aspartate aminotransferase; \ SI = \textit{Le Système International d'Unités} \\ (International System of Units).$ 

### 17.0 CHANGES IN AMENDMENT 1 OF THE STATISTICAL ANALYSIS PLAN

Rationale: This SAP, Amendment 1 is being updated prior to database lock to allow for the non-inflammatory lesion count assessment to be considered as a secondary efficacy endpoint. It will be included in the hierarchy of testing of the secondary endpoints to maintain type 1 error control at 0.05. Since this change is occurring after the completion of all patients in the study, and given that there is no impact on patient safety or study conduct, the protocol will not be amended to reflect this change.

Summary of changes: Sections 10.2, 11.5.1, and 16.2 have been updated to add non-inflammatory lesion count changes from baseline as a secondary efficacy endpoint and to reflect the dual nature of this parameter as being evaluated both for efficacy and for safety.

#### 18.0 REFERENCES

Kim, Y, Won S; Adjusted proportion difference and confidence interval in stratified randomized trials. PharmaSUG Proceedings. 2013;SP04.

Littell, R. C., Milliken, G. A., Stroup, W. W., Wolfinger, R. D., and Schabenberger, O. (2006), *SAS for Mixed Models*, Second Edition, Cary, NC: SAS Press.

O'Kelly M, Ratitch B. Clinical trials with missing data: a guide for practioner. John Wiley & Sons 2014.

Rubin, DB. Inference and missing data. Biometrika. 1976;63:581-592.

Rubin, DB. Multiple imputation for nonresponse in surveys. John Wiley & Sons 1987.

Rubin, DB. Multiple imputation after 18+ Years. J. of the Amer Statistical Assoc. 1996;91: 473-489.

Wilson, EB, Hilferty, MM. The distribution of chi-squared. Proceedings of the National Academy of Sciences, Washington. 1931;17:12,684–688.

US Census Bureau. US Department of Commerce Economics and Statistics Administration US Census Bureau. Census Regions and Divisions of the United States. 2013 Apr 17. Available from: http://www2.census.gov/geo/pdfs/maps-data/maps/reference/us regdiv.pdf. Accessed 2015 Oct 06.

Yan, X, Su, XG; Stratified Wilson and Newcombe confidence intervals for multiple binomial proportions. Statistics in Biopharmaceutical Research. 2010;2:3,329-335.

#### 19.0 APPENDICES

# APPENDIX 1 CONVENTIONAL US REPORTING OF REFERENCE RANGES FOR CLINICAL LABORATORY EVALUATIONS



















Special Chemistry Final 30Sect2014 Created by:



### **ALLERGAN**

### 16.1.9 Analysis Plan Prior to Database Lock Study SC1401

| Date (DD/MMM/YYYY)/Time (PT) | Signed by: | Justification |
|------------------------------|------------|-------------------------------|
| 03-Mar-2017 13:31 GMT-080 | | Biostatistics Approval |
| 03-Mar-2017 13:45 GMT-080 | | Clinical Development Approval |
| 03-Mar-2017 14:18 GMT-080 | | Biostatistics Approval |
| 03-Mar-2017 15:00 GMT-080 | | Biostatistics Approval |

| SMQ | Sub-SMQ | Scope | Preferrerd Term Name |
|---|---|---|---|
| Gastrointestinal | Gastrointestinal | Narrow | Acid peptic disease |
| nonspecific | nonspecific | Narrow | Duodenogastric reflux |
| inflammation | dysfunction (SMQ) | Narrow | Dyspepsia |
| and | | Narrow | Gastrooesophageal reflux disease |
| dysfunctional | | Narrow | Gastrooesophageal sphincter insufficiency |
| conditions | Gastrointestinal | Narrow | Colitis |
| (SMQ) | nonspecific | Narrow | Duodenitis |
| | inflammation (SMQ) | Narrow | Enteritis |
| | | Narrow | Erosive duodenitis |
| | | Narrow | Erosive oesophagitis |
| | | Narrow | Feline oesophagus |
| | | Narrow | Functional gastrointestinal disorder |
| | | Narrow | Gastric mucosa erythema |
| | | Narrow | Gastritis |
| | | Narrow | Gastritis erosive |
| | | Narrow | Gastroduodenitis |
| | | Narrow | Gastrointestinal erosion |
| | | Narrow | Gastrointestinal mucosa hyperaemia |
| | | Narrow | Gastrointestinal mucosal exfoliation |
| | | Narrow | Haemorrhagic erosive gastritis |
| | | Narrow | Intestinal angioedema |
| | | Narrow | Oesophageal mucosa erythema |
| | | Narrow | Oesophagitis |
| | | Narrow | Reactive gastropathy |
| | | Narrow | Reflux gastritis |
| | | Narrow | Remnant gastritis |
| | | Narrow | Ulcerative gastritis |
| | | Broad | Gastrointestinal inflammation |
| | | Broad | Oesophageal irritation |
| | Gastrointestinal | Narrow | Abdominal discomfort |
| | nonspecific symptoms | Narrow | Abdominal distension |
| | and therapeutic | Narrow | Abdominal pain |
| | procedures (SMQ) | Narrow | Abdominal pain lower |
| | | Narrow | Abdominal pain upper |
| | | Narrow | Abdominal symptom |
| | | Narrow | Abdominal tenderness |
| | | Narrow | Abnormal faeces |
| | | Narrow | Aerophagia |
| | | Narrow | Anorectal discomfort |

| SMQ | Sub-SMQ | Scope | Preferrerd Term Name |
|---|---|---|---|
| | | Narrow | Bowel movement irregularity |
| | | Narrow | Change of bowel habit |
| | | Narrow | Constipation |
| | | Narrow | Defaecation urgency |
| | | Narrow | Diarrhoea |
| | | Narrow | Epigastric discomfort |
| | | Narrow | Eructation |
| | | Narrow | Faecal volume decreased |
| | | Narrow | Faecal volume increased |
| | | Narrow | Faeces hard |
| | | Narrow | Faeces soft |
| | | Narrow | Flatulence |
| | | Narrow | Frequent bowel movements |
| | | Narrow | Gastrointestinal pain |
| | | Narrow | Gastrointestinal sounds abnormal |
| | | Narrow | Gastrointestinal toxicity |
| | | Narrow | Infrequent bowel movements |
| | | Narrow | Nausea |
| | | Narrow | Non-cardiac chest pain |
| | | Narrow | Oesophageal discomfort |
| | | Narrow | Oesophageal pain |
| | | Narrow | Vomiting |
| | | Broad | Dysphagia |
| | | Broad | Gastrointestinal tract irritation |
| | | Broad | Regurgitation |
| | | Broad | Retching |
| | | Broad | Steatorrhoea |
| | | Broad | Vomiting projectile |
| Gastrointestinal | Gastrointestinal | Narrow | Anal haemorrhage |
| perforation, | haemorrhage (SMQ) | Narrow | Anal ulcer haemorrhage |
| ulceration, | | Narrow | Anastomotic haemorrhage |
| haemorrhage or | | Narrow | Anastomotic ulcer haemorrhage |
| obstruction | | Narrow | Anorectal varices haemorrhage |
| (SMQ) | | Narrow | Chronic gastrointestinal bleeding |
| | | Narrow | Colonic haematoma |
| | | Narrow | Diarrhoea haemorrhagic |
| | | Narrow | Diverticulitis intestinal haemorrhagic |
| | | Narrow | Diverticulum intestinal haemorrhagic |
| | | Narrow | Duodenal operation |

| SMQ | Sub-SMQ | Scope | Preferrerd Term Name |
|-----|---------|--------|--------------------------------------------|
| | | Narrow | Duodenal ulcer haemorrhage |
| | | Narrow | Duodenal vascular ectasia |
| | | Narrow | Duodenitis haemorrhagic |
| | | Narrow | Enterocolitis haemorrhagic |
| | | Narrow | Gastric antral vascular ectasia |
| | | Narrow | Gastric haemangioma |
| | | Narrow | Gastric haemorrhage |
| | | Narrow | Gastric occult blood positive |
| | | Narrow | Gastric ulcer haemorrhage |
| | | Narrow | Gastric ulcer haemorrhage, obstructive |
| | | Narrow | Gastric varices haemorrhage |
| | | Narrow | Gastritis alcoholic haemorrhagic |
| | | Narrow | Gastritis haemorrhagic |
| | | Narrow | Gastroduodenal haemorrhage |
| | | Narrow | Gastroduodenitis haemorrhagic |
| | | Narrow | Gastrointestinal anastomotic leak |
| | | Narrow | Gastrointestinal angiectasia |
| | | Narrow | Gastrointestinal angiodysplasia haemorrhag |
| | | Narrow | Gastrointestinal haemorrhage |
| | | Narrow | Gastrointestinal polyp haemorrhage |
| | | Narrow | Gastrointestinal ulcer haemorrhage |
| | | Narrow | Haematemesis |
| | | Narrow | Haematochezia |
| | | Narrow | Haemorrhagic erosive gastritis |
| | | Narrow | Haemorrhoidal haemorrhage |
| | | Narrow | Intestinal haematoma |
| | | Narrow | Intestinal haemorrhage |
| | | Narrow | Intestinal varices haemorrhage |
| | | Narrow | Large intestinal haemorrhage |
| | | Narrow | Large intestinal ulcer haemorrhage |
| | | Narrow | Lower gastrointestinal haemorrhage |
| | | Narrow | Mallory-Weiss syndrome |
| | | Narrow | Melaena |
| | | Narrow | Melaena neonatal |
| | | Narrow | Neonatal gastrointestinal haemorrhage |
| | | Narrow | Occult blood positive |
| | | Narrow | Oesophageal haemorrhage |
| | | Narrow | Oesophageal intramural haematoma |
| | | Narrow | Oesophageal ulcer haemorrhage |

| SMQ | Sub-SMQ | Scope | Preferrerd Term Name |
|-----|-------------------|--------|-----------------------------------------|
| | | Narrow | Oesophageal varices haemorrhage |
| | | Narrow | Oesophagitis haemorrhagic |
| | | Narrow | Peptic ulcer haemorrhage |
| | | Narrow | Proctitis haemorrhagic |
| | | Narrow | Rectal haemorrhage |
| | | Narrow | Rectal ulcer haemorrhage |
| | | Narrow | Small intestinal haemorrhage |
| | | Narrow | Small intestinal ulcer haemorrhage |
| | | Narrow | Ulcer haemorrhage |
| | | Narrow | Upper gastrointestinal haemorrhage |
| | | Narrow | White nipple sign |
| | Gastrointestinal | Narrow | Anal dilation procedure |
| | obstruction (SMQ) | Narrow | Anal stenosis |
| | | Narrow | Anastomotic stenosis |
| | | Narrow | Anastomotic ulcer, obstructive |
| | | Narrow | Anorectal stenosis |
| | | Narrow | Appendicolith |
| | | Narrow | Barium impaction |
| | | Narrow | Distal intestinal obstruction syndrome |
| | | Narrow | Duodenal obstruction |
| | | Narrow | Duodenal stenosis |
| | | Narrow | Duodenal ulcer perforation, obstructive |
| | | Narrow | Duodenal ulcer, obstructive |
| | | Narrow | Fibrosing colonopathy |
| | | Narrow | Fixed bowel loop |
| | | Narrow | Gallstone ileus |
| | | Narrow | Gastric ileus |
| | | Narrow | Gastric stenosis |
| | | Narrow | Gastric stent insertion |
| | | Narrow | Gastric ulcer haemorrhage, obstructive |
| | | Narrow | Gastric ulcer perforation, obstructive |
| | | Narrow | Gastric ulcer, obstructive |
| | | Narrow | Gastric volvulus |
| | | Narrow | Gastrointestinal anastomotic leak |
| | | Narrow | Gastrointestinal dilation procedure |
| | | Narrow | Gastrointestinal motility disorder |
| | | Narrow | Gastrointestinal obstruction |
| | | Narrow | Gastrointestinal stenosis |
| | | Narrow | Ileal stenosis |

| SMQ | Sub-SMQ | Scope | Preferrerd Term Name |
|-----|---------|--------|----------------------------------------|
| | | Narrow | Ileus |
| | | Narrow | Ileus paralytic |
| | | Narrow | Ileus spastic |
| | | Narrow | Impaired gastric emptying |
| | | Narrow | Intestinal fibrosis |
| | | Narrow | Intestinal malrotation repair |
| | | Narrow | Intestinal obstruction |
| | | Narrow | Intestinal scarring |
| | | Narrow | Intestinal stenosis |
| | | Narrow | Intussusception |
| | | Narrow | Jejunal stenosis |
| | | Narrow | Large intestinal obstruction |
| | | Narrow | Large intestinal obstruction reduction |
| | | Narrow | Large intestinal stenosis |
| | | Narrow | Malignant bowel obstruction |
| | | Narrow | Mechanical ileus |
| | | Narrow | Necrotising colitis |
| | | Narrow | Necrotising gastritis |
| | | Narrow | Necrotising oesophagitis |
| | | Narrow | Neonatal intestinal obstruction |
| | | Narrow | Obstruction gastric |
| | | Narrow | Obstructive defaecation |
| | | Narrow | Oesophageal compression |
| | | Narrow | Oesophageal dilation procedure |
| | | Narrow | Oesophageal obstruction |
| | | Narrow | Oesophageal stenosis |
| | | Narrow | Peptic ulcer perforation, obstructive |
| | | Narrow | Peptic ulcer, obstructive |
| | | Narrow | Postoperative ileus |
| | | Narrow | Prepyloric stenosis |
| | | Narrow | Pylorus dilation procedure |
| | | Narrow | Rectal obstruction |
| | | Narrow | Rectal stenosis |
| | | Narrow | Small intestinal obstruction |
| | | Narrow | Small intestinal obstruction reduction |
| | | Narrow | Small intestinal stenosis |
| | | Narrow | Stomach dilation procedure |
| | | Narrow | Stricturoplasty |
| | | Narrow | Subileus |

| SMQ | Sub-SMQ | Scope | Preferrerd Term Name |
|-----|-------------------|--------|-----------------------------------------|
| | | Narrow | Volvulus |
| | | Narrow | Volvulus repair |
| | Gastrointestinal | Narrow | Abdominal abscess |
| | perforation (SMQ) | Narrow | Abdominal hernia perforation |
| | | Narrow | Abdominal wall abscess |
| | | Narrow | Abscess intestinal |
| | | Narrow | Acquired tracheo-oesophageal fistula |
| | | Narrow | Anal abscess |
| | | Narrow | Anal fistula |
| | | Narrow | Anal fistula excision |
| | | Narrow | Anal fistula infection |
| | | Narrow | Anastomotic ulcer perforation |
| | | Narrow | Anovulvar fistula |
| | | Narrow | Aorto-duodenal fistula |
| | | Narrow | Aorto-oesophageal fistula |
| | | Narrow | Appendiceal abscess |
| | | Narrow | Appendicitis perforated |
| | | Narrow | Arterioenteric fistula |
| | | Narrow | Atrio-oesophageal fistula |
| | | Narrow | Chemical peritonitis |
| | | Narrow | Colon fistula repair |
| | | Narrow | Colonic abscess |
| | | Narrow | Colonic fistula |
| | | Narrow | Diverticular fistula |
| | | Narrow | Diverticular perforation |
| | | Narrow | Douglas' abscess |
| | | Narrow | Duodenal perforation |
| | | Narrow | Duodenal ulcer perforation |
| | | Narrow | Duodenal ulcer perforation, obstructive |
| | | Narrow | Duodenal ulcer repair |
| | | Narrow | Enterocolonic fistula |
| | | Narrow | Enterocutaneous fistula |
| | | Narrow | Enterovesical fistula |
| | | Narrow | Fistula of small intestine |
| | | Narrow | Gastric fistula |
| | | Narrow | Gastric fistula repair |
| | | Narrow | Gastric perforation |
| | | Narrow | Gastric ulcer perforation |
| | | Narrow | Gastric ulcer perforation, obstructive |

| SMQ | Sub-SMQ | Scope | Preferrerd Term Name |
|-----|---------|--------|---------------------------------------|
| | | Narrow | Gastrointestinal anastomotic leak |
| | | Narrow | Gastrointestinal fistula |
| | | Narrow | Gastrointestinal fistula repair |
| | | Narrow | Gastrointestinal perforation |
| | | Narrow | Gastrointestinal ulcer perforation |
| | | Narrow | Gastropleural fistula |
| | | Narrow | Gastrosplenic fistula |
| | | Narrow | Ileal perforation |
| | | Narrow | Ileal ulcer perforation |
| | | Narrow | Inguinal hernia perforation |
| | | Narrow | Intestinal fistula |
| | | Narrow | Intestinal fistula infection |
| | | Narrow | Intestinal fistula repair |
| | | Narrow | Intestinal perforation |
| | | Narrow | Intestinal ulcer perforation |
| | | Narrow | Jejunal perforation |
| | | Narrow | Jejunal ulcer perforation |
| | | Narrow | Large intestinal ulcer perforation |
| | | Narrow | Large intestine perforation |
| | | Narrow | Lower gastrointestinal perforation |
| | | Narrow | Mesenteric abscess |
| | | Narrow | Neonatal intestinal perforation |
| | | Narrow | Oesophageal fistula |
| | | Narrow | Oesophageal fistula repair |
| | | Narrow | Oesophageal perforation |
| | | Narrow | Oesophageal rupture |
| | | Narrow | Oesophageal ulcer perforation |
| | | Narrow | Oesophagobronchial fistula |
| | | Narrow | Oesophagopleural fistula |
| | | Narrow | Paraoesophageal abscess |
| | | Narrow | Peptic ulcer perforation |
| | | Narrow | Peptic ulcer perforation, obstructive |
| | | Narrow | Perforated peptic ulcer oversewing |
| | | Narrow | Perforated ulcer |
| | | Narrow | Perineal abscess |
| | | Narrow | Perirectal abscess |
| | | Narrow | Peritoneal abscess |
| | | Narrow | Peritonitis |
| | | Narrow | Peritonitis bacterial |

| SMQ | Sub-SMQ | Scope | Preferrerd Term Name |
|-----|---------------------|--------|---------------------------------------|
| | | Narrow | Procedural intestinal perforation |
| | | Narrow | Rectal abscess |
| | | Narrow | Rectal fistula repair |
| | | Narrow | Rectal perforation |
| | | Narrow | Rectoprostatic fistula |
| | | Narrow | Rectourethral fistula |
| | | Narrow | Retroperitoneal abscess |
| | | Narrow | Small intestinal perforation |
| | | Narrow | Small intestinal ulcer perforation |
| | | Narrow | Umbilical hernia perforation |
| | | Narrow | Upper gastrointestinal perforation |
| | Gastrointestinal | Narrow | Bloody peritoneal effluent |
| | perforation, ulcer, | Narrow | Corrosive gastritis |
| | haemorrhage, | Narrow | Fixed bowel loop |
| | obstruction non- | Narrow | Gastric atony |
| | specific | Narrow | Gastric hypomotility |
| | findings/procedures | Narrow | Gastrointestinal hypomotility |
| | (SMQ) | Narrow | Haemorrhagic ascites |
| | | Narrow | Intra-abdominal haematoma |
| | | Narrow | Intra-abdominal haemorrhage |
| | | Narrow | Megacolon |
| | | Narrow | Mesenteric haematoma |
| | | Narrow | Mesenteric haemorrhage |
| | | Narrow | Mucosal erosion |
| | | Narrow | Mucosal haemorrhage |
| | | Narrow | Mucosal ulceration |
| | | Narrow | Narcotic bowel syndrome |
| | | Narrow | Oesophageal achalasia |
| | | Narrow | Oesophageal atony |
| | | Narrow | Oesophageal hypomotility |
| | | Narrow | Peritoneal haematoma |
| | | Narrow | Peritoneal haemorrhage |
| | | Narrow | Retroperitoneal haematoma |
| | | Narrow | Retroperitoneal haemorrhage |
| | | Narrow | Toxic dilatation of intestine |
| | Gastrointestinal | Narrow | Acute haemorrhagic ulcerative colitis |
| | ulceration (SMQ) | Narrow | Anal erosion |
| | | Narrow | Anal ulcer |
| | | Narrow | Anal ulcer haemorrhage |

| SMQ | Sub-SMQ | Scope | Preferrerd Term Name |
|-----|---------|--------|----------------------------------------|
| | | Narrow | Anastomotic ulcer |
| | | Narrow | Anastomotic ulcer haemorrhage |
| | | Narrow | Anastomotic ulcer perforation |
| | | Narrow | Anorectal ulcer |
| | | Narrow | Colitis erosive |
| | | Narrow | Colitis ulcerative |
| | | Narrow | Cytomegalovirus gastrointestinal ulcer |
| | | Narrow | Duodenal ulcer |
| | | Narrow | Duodenal ulcer haemorrhage |
| | | Narrow | Duodenal ulcer perforation |
| | | Narrow | Duodenal ulcer repair |
| | | Narrow | Duodenal ulcer, obstructive |
| | | Narrow | Erosive duodenitis |
| | | Narrow | Erosive oesophagitis |
| | | Narrow | Gastric ulcer |
| | | Narrow | Gastric ulcer haemorrhage |
| | | Narrow | Gastric ulcer haemorrhage, obstructive |
| | | Narrow | Gastric ulcer helicobacter |
| | | Narrow | Gastric ulcer perforation |
| | | Narrow | Gastric ulcer perforation, obstructive |
| | | Narrow | Gastric ulcer surgery |
| | | Narrow | Gastritis erosive |
| | | Narrow | Gastritis haemorrhagic |
| | | Narrow | Gastritis hypertrophic |
| | | Narrow | Gastroduodenal ulcer |
| | | Narrow | Gastrointestinal anastomotic leak |
| | | Narrow | Gastrointestinal erosion |
| | | Narrow | Gastrointestinal ulcer |
| | | Narrow | Gastrointestinal ulcer haemorrhage |
| | | Narrow | Gastrointestinal ulcer management |
| | | Narrow | Gastrointestinal ulcer perforation |
| | | Narrow | Haemorrhagic erosive gastritis |
| | | Narrow | Ileal ulcer |
| | | Narrow | Ileal ulcer perforation |
| | | Narrow | Intestinal scarring |
| | | Narrow | Intestinal ulcer |
| | | Narrow | Intestinal ulcer perforation |
| | | Narrow | Ischaemic ulcer |
| | | Narrow | Jejunal ulcer |

# Study SC1401 Appendix 16.1.9.2 Page 10 of 10 Pre-Specified Preferred Terms Used for Gastrointestinal Standardised MedDRA Queries

| SMQ | Sub-SMQ | Scope | Preferrerd Term Name |
|-----|---------|--------|--------------------------------------------|
| | | Narrow | Jejunal ulcer perforation |
| | | Narrow | Large intestinal ulcer |
| | | Narrow | Large intestinal ulcer haemorrhage |
| | | Narrow | Large intestinal ulcer perforation |
| | | Narrow | Large intestine erosion |
| | | Narrow | Lip erosion |
| | | Narrow | Necrotising colitis |
| | | Narrow | Necrotising gastritis |
| | | Narrow | Necrotising oesophagitis |
| | | Narrow | Oesophageal ulcer |
| | | Narrow | Oesophageal ulcer haemorrhage |
| | | Narrow | Oesophageal ulcer perforation |
| | | Narrow | Oesophagitis ulcerative |
| | | Narrow | Peptic ulcer |
| | | Narrow | Peptic ulcer haemorrhage |
| | | Narrow | Peptic ulcer helicobacter |
| | | Narrow | Peptic ulcer perforation |
| | | Narrow | Peptic ulcer perforation, obstructive |
| | | Narrow | Peptic ulcer, obstructive |
| | | Narrow | Perforated peptic ulcer oversewing |
| | | Narrow | Perforated ulcer |
| | | Narrow | Proctitis ulcerative |
| | | Narrow | Prophylaxis against gastrointestinal ulcer |
| | | Narrow | Rectal ulcer |
| | | Narrow | Rectal ulcer haemorrhage |
| | | Narrow | Small intestinal ulcer haemorrhage |
| | | Narrow | Small intestinal ulcer perforation |
| | | Narrow | Small intestine ulcer |
| | | Narrow | Stress ulcer |
| | | Narrow | Ulcer |
| | | Narrow | Ulcer haemorrhage |
| | | Narrow | Ulcerative gastritis |